CLINICAL TRIAL: NCT05537363
Title: The Effects of an Agility Training and Its Relation to Motor, Cognitive Performance and Fall Risk in Elderly Adults With and Without Mild Cognitive Impairment
Brief Title: Agility Training and Its Relations in Elderly Adults With and Without MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202112236RINB
Record Dates: First submitted 2022-07-24; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-05

CONDITIONS: Elderly Adults; Mild Cognitive Impairment; Healthy
Keywords: Aging; Agility training; Cognition function; Fall; Mild Cognitive Impairment; Motor function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Healthy adults (No Intervention): Year 1: To assess levels of agility and agility performance in relation to the motor and cognitive abilities of healthy young adults, healthy elderly, and elderly with MCI.
- Healthy elderly and mild cognitive impairment elderly (No Intervention): Year 1: To assess levels of agility and agility performance in relation to the motor and cognitive abilities of healthy young adults, healthy elderly, and elderly with MCI.
- Mild cognitive impairment elderly with health education (Active Comparator): Year 2: To determine the short and long-term effects of a multicomponent training protocol and an agility training protocol on agility, motor, and cognitive function in elderly with MCI.
  Interventions: Other: Health education
- Mild cognitive impairment elderly with multicomponent training (Experimental): Year 2: To determine the short and long-term effects of a multicomponent training protocol and an agility training protocol on agility, motor, and cognitive function in elderly with MCI.
  Interventions: Other: Multicomponent training
- Mild cognitive impairment elderly with agility training (Experimental): Year 2: To determine the short and long-term effects of a multicomponent training protocol and an agility training protocol on agility, motor, and cognitive function in elderly with MCI.
  Interventions: Other: Agility training
- Healthy elderly with health education (Active Comparator): Year 3: To determine the short and long-term effects of a multicomponent training protocol and an agility training protocol on agility ability, motor, and cognitive function in healthy elderly adults.
  Interventions: Other: Health education
- Healthy elderly with multicomponent training (Experimental): Year 3: To determine the short and long-term effects of a multicomponent training protocol and an agility training protocol on agility ability, motor, and cognitive function in healthy elderly adults.
  Interventions: Other: Multicomponent training
- Healthy elderly with agility training (Experimental): Year 3: To determine the short and long-term effects of a multicomponent training protocol and an agility training protocol on agility ability, motor, and cognitive function in healthy elderly adults.
  Interventions: Other: Agility training

INTERVENTIONS:
Other: Health education — Participants in the control group will receive health educational guidelines. Guideline contents include home-based exercise program, nutrition recommendations, and fall prevention education.
  Arms: Healthy elderly with health education; Mild cognitive impairment elderly with health education
Other: Multicomponent training — Multicomponent exercises will be designed according to the results of Part I of our study. Results of Part I of this study will determine the contributing factors of agility, such as muscle strength, endurance, and cognitive function. A physical therapist will train the participants 3-4 exercises (3-4 factors) in each session. The physical therapist will adjust the difficulty of each exercise according to the participant's ability and condition.
  Arms: Healthy elderly with multicomponent training; Mild cognitive impairment elderly with multicomponent training
Other: Agility training — The agility-based task-specific exercises will be conducted in this group and will incorporate stop-and-go, change in direction, change in velocity, acceleration and deceleration training. There are four training configurations with 3 levels of difficulty, which will be manipulated by increasing speed, distance, number of repetitions, number of directions, congruency, and/or complexity of the task, or by decreasing the number and duration of the rest intervals. The physical therapist will adjust the difficulty of each exercise according to the participant's ability and condition.
  Arms: Healthy elderly with agility training; Mild cognitive impairment elderly with agility training

SUMMARY:
The following three-part proposal will focus on the effects of agility training as well as the relationship between agility ability and motor and cognitive function, and risk of falls in elderly adults with or without mild cognitive impairment (MCI).

Part I is a cross-sectional study design that will assess the level of agility in healthy young adults, healthy elderly adults, and elderly adults with MCI to determine the effect of aging and cognition decline on agility and the relations between agility, cognitive, and motor functions. Thirty participants will be screened for eligibility and recruited for each group (90 participants total). After collecting basic data, all participants will undergo cognitive and motor function tests, as well as an agility test. Cognitive function tests include tests of global cognition, working memory, mental set shifting, and selective attention. Motor function tests include tests of single and dual task walking, strength, power, balance, flexibility, and endurance. The agility test contains stop-and-go, change of direction, and spatial orientation components. Functional near-infrared spectroscopy (fNIRS) will be used to evaluate the brain activation during the agility test, cognitive tests, and single and dual task walking. Results from all tests will be used to determine the motor, cognitive, and other predictive factors associated with agility performance, and will be used in the design of the training program in Part II and III.

Part II and III are single-blinded randomized controlled trials that will explore the short and long-term effects of a multicomponent training and an agility training protocol on agility, motor, and cognitive function in elderly adults with and without MCI. Seventy-five elderly adults with MCI (Part II) and seventy-five healthy elderly (Part III) will be recruited. After screening for eligibility and collection of demographic data, participants will undergo a pretest assessment. In addition to the motor, cognitive, and agility tests used in Part I, information on history of falls, falls efficacy, and quality of life will be assessed for each participant. Brain activation will be assessed during the agility test, cognitive tests, and single and dual task walking assessments using fNIRS. Participants will be randomly allocated into one of three groups: the control group, the multicomponent training group, or the agility training group (n=25 in each group). Intervention will be executed at a frequency of 45 minutes per session, 2 times a week for 8 weeks. The control group will receive home-based health education guidelines. The multicomponent training group will engage in 3 to 4 exercises each training session comprising the influencing factors of agility, and the agility training group will engage in integrated task-specific training. A post-test will be conducted after the 8-week intervention, and 1-month, 6-month, and 12-month follow-ups will be conducted for elderly adults with MCI. The healthy elderly adults will be assessed after the intervention and at the 1-month follow-up after training.

ELIGIBILITY:
Part 1:

Inclusion Criteria:

1. has a score of ≥ 24 on the Mini-Mental State Examination (MMSE)
2. able to walk independently for more than 30 meters without assistive aids
3. able to follow orders

Exclusion Criteria:

1. poorly-controlled or unstable systematic disease
2. has a history of central nervous system disease
3. currently taking antidepressants, anti-anxiety, or other psychiatric drugs that may affect blood flow in the brain
4. subjects with achromatopsia

Part 2:

Inclusion Criteria:

1. older than 65 years old
2. score of Mini-Mental State Examination (MMSE) ≥ 24 and score of Montreal Cognitive Assessment (MoCA) ≤ 26
3. able to walk independently for more than 30 meters without assistive aids
4. able to follow orders

Exclusion Criteria:

1. poorly controlled or unstable systematic disease
2. has a history of central nervous system disease
3. currently taking antidepressants, anti-anxiety, or other psychiatric drugs that may affect blood flow in the brain
4. has other medical conditions for which exercise is contraindicated
5. subjects with achromatopsia

Part 3:

Inclusion Criteria:

1. older than 65 years old
2. score of Mini-Mental State Examination (MMSE) ≥ 24
3. able to walk independently for more than 30 meters without assistive aids
4. able to follow orders

Exclusion Criteria:

1. poorly controlled or unstable systematic disease
2. has a history of central nervous system disease
3. currently taking antidepressants, anti-anxiety, or other psychiatric drugs that may affect blood flow in the brain
4. has other medical conditions for which exercise is contraindicated
5. subjects with achromatopsia

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Agility Challenge for the Elderly (ACE) | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  An agility course developed for a 9m x 18m volleyball court and includes three segments that each aim to test a specific aspect of agility, including stop-and-go, change of direction, and spatial orientation.

SECONDARY OUTCOMES:
Fall history and fear of falls | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  Fall history will be recorded by the number of fall episodes in the past 6 months and whether it caused injury.
Quality of life (QOL) | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  Quality of life (QOL) will be evaluated by Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36).
Brain activation | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  A multichannel wearable fNIRS imaging system (NIRSport2, NIRx Medical Technologies LLC, Glen Head, NY, USA) will be used to detect the hemodynamics of brain areas associated with the agility test, cognitive tasks, and single and dual task walking test.
Montreal Cognitive Assessment (MoCA) | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  MoCA contains 16 items and 11 categories to assess multiple cognitive domains, is a screening instrument for MCI, and its validity has been established in various clinical groups and countries.
Mental set shifting | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  The Wisconsin Card Sorting Test (WCST) will be used to measure participants' ability to shift their cognitive ability in response to the demands of environment.
Working memory | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  The backward digit span test (DGS) will be used to measure working memory.
Selective attention and inhibition | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  The Stroop Color and Word Test (SCWT) will be used to measure selective attention.
Motor Function | Part 1:Baseline; Part 2: Pre-intervention, 8 weeks, 12 weeks, 8-month, and 14-month
  Walking performance, normal walking, cognitive dual-task walking, muscle strength of bilateral lower limbs, five times sit to stand test, timed up and go, quiet static standing task, and the 360° turning task, flexibility, 6-minute walk test (6WMT).

CONTACTS AND LOCATIONS:
Overall Officials: Yan Ci Liu, PhD, Principal Investigator — National Taiwan University